CLINICAL TRIAL: NCT05609773
Title: Comparing Intubation Rates in the Delivery Room by Interface
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Illinois College of Medicine at Peoria (Other)
Collaborators: Children's Hospital of Illinois (Unknown); OSF Healthcare System (Other)
Responsible Party: Sponsor
Other Study IDs: 1783154
Record Dates: First submitted 2022-10-31; First posted 2022-11-08 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Ventilator Lung; Newborn
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although the majority of premature neonates < 30 weeks gestion require positive pressure ventilation (PPV) at birth, the optimal interface to provide PPV has not been determined. Preferably this support would be provided by non-invasive means to prevent the development of bronchopulmonary dysplasia. Resuscitation with a face mask, single nasal tube, nasal prongs, and/or LMA are all approved methods of resuscitation per NRP as of 2010. Face masks have been associated with more dead space, air leak and airway obstruction however are the most commonly used interface. Recently, the Trigeminal Cardiac Reflex has been described, which can be induced with the placement of a facemask, resulting in bradycardia and apnea. Bi-nasal prongs (RAM cannula) have been found in studies to be associated with lower intubation rates in the delivery room (down to 24 weeks gestation), less need for epinephrine, chest compressions, and subsequent invasive ventilation. In addition to the potential practical advantages of bi-nasal prong resuscitation, there is evidence to suggest that ventilation through the nose may stimulate the subepithelial receptors of the upper airways causing an increase in respiratory rate and depth.

ELIGIBILITY:
Inclusion Criteria:

All resuscitated infants < 30 weeks' gestation born at OSF SFMC

Exclusion Criteria:

Diagnosis of congenital diaphragmatic hernia No PPV needed, or no resuscitation desired due to major congenital anomalies or peri- viable status

Ages: 0 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All resuscitated infants < 30 weeks' gestation born at OSF SFMC.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Comparing Intubation Rates in the Delivery Room by Interface | 3 years
  We hypothesize that there will be at least a 40% reduction in the rate of intubation for patients born < 30 weeks' gestation when bi-nasal prongs are utilized for neonatal resuscitation vs face mask.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Fischer, MD, Principal Investigator — University of Illinois College of Medicine at Peoria
Locations (1):
- University of Illinois College of Medicince, Peoria, Illinois, United States

DOCUMENTS (1):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT05609773/Prot_001.pdf